CLINICAL TRIAL: NCT05822206
Title: Development of a Trauma Informed Intervention to Support Adaptive Engagement in Care Among MSM Living With HIV: Project THRIVE+
Brief Title: Trauma Informed Intervention to Support Engagement in HIV Care Among MSM (THRIVE+)
Acronym: THRIVE+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Fenway Institute (Other); Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Conall O'Cleirigh, Director of Behavioral Medicine Program, Department of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 931482-1
Record Dates: First submitted 2020-06-26; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: HIV/AIDS; Trauma
Keywords: MSM; HIV/AIDS; Trauma; Engagement in care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participants are randomized into one of two conditions: treatment (Cognitive Behavioral Therapy for Trauma and Self-Care; CBT-TSC) or control. The CBT-TSC condition consists of 10 therapy sessions and 3 follow-up visits. The control condition consists of 2 therapy sessions and 3 follow-up visits. The first two therapy sessions, which are received by all participants regardless of condition, employ LifeSteps and sexual decision making techniques. The remaining eight therapy sessions, which only those in the CBT-TSC condition receive, address thoughts and behaviors associated with trauma distress and poor engagement in HIV care.
Who Masked: Outcomes Assessor
Masking Description: Randomization is known to the study investigator, study clinician, project coordinator, and participant. The outcomes assessor is privy to randomization information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants in the Treatment arm receive 2 therapy sessions on LifeSteps and sexual decision-making, as well at 8 sessions of Cognitive Behavioral Therapy for Trauma and Self-Care (CBT-TSC). Participants then participate in 3-, 6-, and 9-month follow-up assessments.
  Interventions: Behavioral: CBT-TSC; Behavioral: Life Steps and Sexual Decision-Making
- Control (Other): Participants in the Control arm receive 2 therapy sessions on LifeSteps and sexual decision-making. Participants then participate in 3-, 6-, and 9-month follow-up assessments.
  Interventions: Behavioral: Life Steps and Sexual Decision-Making

INTERVENTIONS:
Behavioral: CBT-TSC — Cognitive Behavioral Therapy for Trauma and Self-Care
  Arms: Treatment
Behavioral: Life Steps and Sexual Decision-Making

SUMMARY:
This purpose of this project is to specify and provide an initial test of a 10 session, individual-based cognitive therapy intervention to address symptoms of PTSD and poor engagement in HIV care among men who have sex with men (MSM) with trauma histories

DETAILED DESCRIPTION:
The proposed intervention will incorporate the most current approaches to mediating trauma responses and stressors related to experiences of HIV stigma and homonegativity with cognitive-processing therapy, an empirically validated, cognitive-behavioral intervention for reducing negative consequences of traumatic stress. This intervention intends to improve uptake of HIV care in the prevention, engagement, and care cascade while also addressing the mental health needs of HIV-positive persons in a program of research that leads to outcomes in the short-term. If found to be efficacious, this intervention can also be scalable across clinical settings.

The study will be implemented at The Fenway Institute at Fenway Health (TFI) and at Ryerson University, Toronto, Canada and Drs. O'Cleirigh and Hart will assume the responsibility of coordinating the study across sites.

Randomization will be to the 10 session intervention or to two medication adherence/engagement in care sessions.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* is a man who has sex with men
* has a history of trauma and is experiencing trauma-related distress (as operationalized by a score of >/= 20 on the Davidson Trauma Scale)
* is sub-optimally engaged in HIV care (as operationalized by missing 1 or more HIV care appointments in the past 12 months, having a detectable viral load at most recent testing, or having poor adherence - </=80% - to HIV medications)

Exclusion Criteria:

* has a significant mental health diagnosis that requires immediate treatment (e.g., acute major depression; panic disorder; any psychotic disorder)
* unable to complete the informed consent process (e.g., substantial cognitive impairment, inadequate English language skills).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — To be eligible for the study, an individual needs to identify as male and have been assigned male at birth.
Enrollment: 40 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
ACTG Adherence Interview | up to 4 times over 9 months
  HIV medication adherence is collected at all major time points (baseline, 3 month follow-up, 6 month follow-up, and 9 month follow-up) via self-report, using the AIDS Clinical Trials Group Adherence Interview. Participants are asked to give the number of doses they take of each of their HIV medications per day, and to note how many doses were missed at 4 time time points (yesterday, day before yesterday, 3 days ago, in the past 2 weeks).

SECONDARY OUTCOMES:
Davidson Trauma Scale | 1 week
  The Davidson Trauma Scale measures the frequency and severity of PTSD symptoms in the past week, and is conducted at each study visit (baseline, weekly visits, and all follow-up visits). Each item on the 17-item scale is scored 0-4 on frequency (0 = not at all; 4 = every day) and severity (0 = not at all distressing; 4 = extremely distressing), yielding a total between 0 and 136.
Viral Load | baseline and 9 months
  Most recent viral load is collected from each participant at baseline (first study visit) and at 9 month follow-up (final study visit) through medical record abstraction.

CONTACTS AND LOCATIONS:
Overall Officials: Conall O'Cleirigh, PhD, Principal Investigator — Fenway Health
Locations (2):
- Fenway Community Health, Boston, Massachusetts, United States
- Ryerson University, Toronto, Ontario, Canada